CLINICAL TRIAL: NCT02436616
Title: Wireless Novel microEEG for Neonatal Apnea and Community Neurological Network
Brief Title: microEEG for Neonatal Apnea, Bradycardia and Desaturation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bio-Signal Group Corp. (Industry)
Collaborators: State University of New York - Downstate Medical Center (Other); Brookdale University Hospital Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 307016-7
Record Dates: First submitted 2014-11-25; First posted 2015-05-07 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2014-11

CONDITIONS: Apnea; Bradycardia; Premature Birth; Seizures
Keywords: EEG; Preterm Infants; Neonate; wireless
MeSH Terms: conditions — Apnea; Bradycardia; Premature Birth; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EEG monitoring: All subjects enrolled in this observational study will undergo EEG monitoring using the microEEG device.
  Interventions: Device: microEEG

INTERVENTIONS:
Device: microEEG — microEEG is a miniature, wireless, and battery-powered EEG device used to obtain EEG recording in challenging environment. All infants have an initial EEG at study enrollment. Follow up microEEGs will be performed at approximately 2-4 week intervals, depending on the Corrected Gestational Age (CGA).
  If ABD events have not resolved at 34 weeks, an 8 hour recording will be performed prior to discharge or at 42 weeks CGA, whichever comes first. EEG will be assessed in 3 hour epochs. The EEG will be reviewed off line by two blinded neurologists and classified as normal or abnormal based on CGA and other findings. Follow up EEGs will be scored similarly, with emphasis on maturation.

SUMMARY:
The study utilizes microEEG (a novel miniaturized, FDA approved EEG device) to prospectively investigate the cerebral electrical activity of infants with Apnea, Bradycardia and Desaturation events. This project will also assess the feasibility of using the microEEG device in the Neonatal Intensive Care Unit (NICU) setting and the feasibility of remote centralized interpretation in this setting.

DETAILED DESCRIPTION:
Most preterm infants have episodes of apnea (cessation of breathing), bradycardia (low heart rate), and desaturations (low levels of oxygen in the blood) (ABD events). The resolution of ABD episodes depends to a large extent on the maturation of the central nervous system (CNS). The electroencephalogram (EEG) is a reliable and noninvasive tool for recording the electrical activity of the CNS. The relationship between ABD events and cerebral electrical activity has not been well investigated. The investigators seek to examine the relationship between EEG findings and the resolution of ABD events in the developing premature infant.

To investigate this relationship and obtain findings which are relevant to clinical care, a variety of obstacles need to be overcome. Among these obstacles is the high cost of standard EEG machines, inability of most standard machines to operate in electrically-noisy environments such as the NICU, and the absence of full-time coverage neurologists for prompt EEG interpretation. The investigators seek to determine the feasibility of obtaining an artifact-free EEG in the NICU with accurate detection of background rhythm abnormalities. The investigators will utilize an existing digital wireless telemetry unit, the "microEEG" for the NICU for this purpose. The microEEG device is specifically designed to overcome obstacles to standard EEG recording.

To address the shortage of trained pediatric neurophysiologists, the investigators will investigate the feasibility of a case management system for centralized EEG interpretation using off-site neurologists.

Finally, the investigators will examine the inter-rater reliability of EEG interpretation in the developing premature infant. This will allow the development of consensus guidelines for EEG interpretations.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age (GA) 24-32 weeks
2. postnatal ages 0-30 days. The patients will be recruited upon manifesting one of the following

   * apneas (cessation of breathing > 10 seconds) x2 in a 12 hour span
   * bradycardias (HR < 100/min) x2 in 12 hours
   * oxygen desaturations (<80%) x 2 in 12 hours
   * a single ABD event that does not resolve with stimulation or an increase in fractional oxygen delivery (FiO2).

Exclusion Criteria:

1. major malformations
2. The infant has exposed dermis on the scalp due to immaturity
3. Any scalp skin lesions such as pustules, large abrasions The patient will be Withdrawn if

   * Informed consent is withdrawn
   * adverse events (i.e..scalp lesions) develop

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature Infants born in hospital at the study centers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between EEG background activity and resolution of Apnea, Bradycardia and Desaturation | Initial 8-9 hours EEG will be done upon study enrollment in the first 30 days of life.
  Primary outcome measure is to assess the background EEG activity in infants with ABD events and determine the relationship between abnormal initial EEG background activity and the resolution of ABD events at 34 weeks Corrected Gestational Age

SECONDARY OUTCOMES:
Rate of seizure activity. | From study enrollement to resolution of ABD events or 42 weeks corrected gesational age, whichever, comes first.
  All EEG recordings will be assessed by a pediatric neurophysiologist for seizure activity using standard clinical criteria. Based on their findings the rate of seizure will be determined.
Feasibility of microEEG recording in the NICU | From study enrollment (first 30 days of life) to resolution of ABD events or 42 weeks gesational age (whichever comes first)
  Assess the ability of neonatal staff to utilize the microEEG to obtain EEG in the NICU. This will be done by measuring the percentage of completed recordings that are interpretable by a pediatric neurophysiologist.
Interrater reliability of neonatal EEG interpretation | From study enrollment (first 30 days of life) to resolution of ABD events or 42 weeks gesational age (whichever comes first)
  Assess the inter-rater reliability of neonatal EEG interpretations using data obtained in the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Ibrahim, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (2):
- United States (2):
  - State University of New York/Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center,, Brooklyn, New York

REFERENCES:
- See also: Abstract from International Chil Neurology Congress — http://icnapedia.org/icnc/index.php/icnc/2014/paper/view/585